CLINICAL TRIAL: NCT02267304
Title: Etude Comparative Monocentrique, randomisée, en Cross Over, en Double Aveugle, Contre Placebo, de l'Action de la Morphine et de la Naloxone Dans un modèle Cognitif de Gestion Des Efforts Physiques
Brief Title: Double Blind Randomized, Monocentric, Cross-over, Placebo-controlled Study to Evaluate the Effect of Morphine and Naloxone on Motivation (MBBAnalgesic)
Acronym: MBBAnalgesic
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Other
Other Study IDs: C13-02; 2013-003487-31 (EudraCT Number)
Record Dates: First submitted 2014-09-24; First posted 2014-10-17 (Estimated); Last update posted 2021-08-26 (Actual); Status verified 2021-08

CONDITIONS: Healthy
Keywords: volunteers
MeSH Terms: interventions — Sodium Chloride; Naloxone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Morphine/placebo/naxolone (Experimental)
  Interventions: Drug: 50 mL of sodium chloride (0,9%); Drug: Morphine 0,05mg/kg; Drug: Naloxone 10mg
- Naxolone/morphine/placebo (Experimental)
  Interventions: Drug: 50 mL of sodium chloride (0,9%); Drug: Morphine 0,05mg/kg; Drug: Naloxone 10mg
- placebo/naxolone/morphine (Experimental)
  Interventions: Drug: 50 mL of sodium chloride (0,9%); Drug: Morphine 0,05mg/kg; Drug: Naloxone 10mg

INTERVENTIONS:
Drug: 50 mL of sodium chloride (0,9%)
Drug: Morphine 0,05mg/kg
Drug: Naloxone 10mg

SUMMARY:
The aim of the current study is to examine the role of the opioïd system on the cognitive parameters of motivation. They are embedded in a conceptual framework of motivation that merges decision-making and reinforcement learning theories. Every action is conceived as path from one state to another. The different states are associated to different values (positive for rewards and negative for punishments), and the different actions to different costs (risk, effort and delay). The tasks are designed such that the sensitivity to the state and action parameters can be inferred by fitting computational models.The primary objective is to characterize the effect of Morphine 0,05mg/kg and Naloxone 10mg on cost accumulation slope, assessed in an effort management task, in which participants are asked to squeeze a hand grip during 30 seconds at varying level of effort in order to win monetary payoff. Secondary objectives are to characterize the effect of Morphine 0,05mg/kg and Naloxone 10mg on other cognitive parameters of motivation (assessed with a motivational battery that includes rating, choice and learning tasks).

ELIGIBILITY:
Inclusion Criteria:

* Man or woman, age ≥ 18 and < 50
* Weight between 50 kg and 90 kg.
* No contraindication to effort
* No evolutive pathology that could interfere with the current study signed consent
* medical insurance ("sécurité sociale")

Exclusion Criteria:

* Age < 18 or > 50
* Smokers
* Person under curatorship, or guardianship, or with civil rights deprivation
* History of neurologic or psychiatric pathology
* Chronic or actual consumption of alcohol, or psychotropic drugs
* pregnancy, breastfeeding
* Woman of childbearing potential without effective contraception
* Liver failure
* Severe Cardiovascular Disorders
* Severe Cerebrovascular Discorders
* Morphine (or Naloxone) hypersensitivity/addiction
* Treatment contraindicated: morphine dérivatives, neuroleptics, barbiturate, benzodiazepine, anxiolytics, hypnotics, antidepressant, antihistamine, antihypertensives, beta blocker, baclofen, thalidomide
* Enzyme inducers, (rifampicine, …)
* Treatment that can interfere with the performance of the subject: beta2 adrenergic agonists, analgesics, corticosteroïds, anti-inflammatory drugs, …

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 37 (Actual)
Dates: Start 2013-10-30 (Actual); Primary Completion 2016-08 (Actual); Study Completion 2016-08-30 (Actual)

PRIMARY OUTCOMES:
Cost Accumulation Slope (AU.) | 15 min after first placebo injection, 15 min after morphine (respectively naloxone) injection
  The primary Outcome measure is the change in this parameter between the placebo condition and the morphine (respectively naloxone) condition.This parameter will be infered from the time spent in a effort period versus a rest period within trials of an effort managing task, for each subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Jean -Christophe Corvol, MCU-PH, Principal Investigator — CIC Neurologie GH Pitié Salpêtrière
Locations (1):
- CIC Neurologie GHPS, Paris, France